CLINICAL TRIAL: NCT07081204
Title: Evaluation of the Prevalence of Temporomandibular Disorders and Lts Association With Tooth Wear Measured Using Digital Methods
Brief Title: Evaluation of Temporomandibular Disorders and Their Association With Tooth Wear Using Digital Methods
Status: Completed | Type: Observational
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Mehmet Gözen, DDS, Konya Necmettin Erbakan Üniversitesi
Other Study IDs: 22023.R1
Record Dates: First submitted 2025-07-05; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Tooth Wear; Occlusal Wear of Teeth; Occlusal Analysis; TMJ; Temporomandibular Disorders (TMD)
Keywords: Digital Dentistry; Temporomandibular Disorders; Tooth Wear
MeSH Terms: conditions — Tooth Wear; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Temporomandibular disorders (TMDs) are considered complex conditions in dental practice due to their multifactorial etiology. Over the years, various diagnostic methods have been introduced; however, the most widely accepted model to explain the complexity of TMD is the biopsychosocial model. The Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) Axis I and Axis II protocol is currently regarded as the gold standard for evaluating TMDs. Today, studies employing the DC/TMD framework are conducted in various populations.

This study aims to assess the prevalence of TMD using updated diagnostic criteria. In addition, it seeks to evaluate the presence of tooth wear-one of the common clinical findings associated with TMD-through digital measurement and visual assessment tools, and to investigate its correlation with TMD. Specifically, the study will examine how changes in occlusal contact points due to bruxism and wear are reflected in functional changes within the temporomandibular joint (TMJ) and the extent of tooth wear. The effects of both mild and severe tooth wear on TMJ health and their potential long-term implications for oral health will also be explored.

The primary objective of this study is to determine the prevalence of TMD in the general population using the DC/TMD Axis I and Axis II protocols and to evaluate the impact of tooth wear-measured via digital intraoral scanners-on TMD. Special attention will be given to how changes in occlusal contact due to bruxism and wear influence stress distribution and adaptive remodeling in TMJ structures. Furthermore, the study aims to compare the effects of mild versus severe tooth wear on joint function, ultimately contributing to the development of early diagnosis and intervention strategies.

Additionally, this study seeks to highlight the effectiveness of digital technologies, such as intraoral scanners and 3D modeling, in evaluating the relationship between tooth wear and TMJ disorders. By doing so, the research aims to enhance the existing literature on the link between tooth wear and TMD and provide evidence-based guidance for clinical practice.

DETAILED DESCRIPTION:
This analytical cross-sectional clinical study was conducted at the Department of Prosthodontics, Faculty of Dentistry, Necmettin Erbakan University between November 2024 and May 2025. The study aimed to investigate the relationship between tooth wear, occlusal contact area, and temporomandibular disorders (TMD) using validated diagnostic and digital tools. Ethical approval was granted by the Non-Invasive Clinical Research Ethics Committee of Necmettin Erbakan University (Approval No: 2024/520; Date: 26.12.2024; ID: 22023.R1). Written informed consent was obtained from all participants in accordance with the Declaration of Helsinki.

Sample size was determined using G*Power software (v3.1), with an effect size of f = 0.33, alpha = 0.05, and power = 0.90, indicating that a minimum of 40 participants per group was required. A total of 120 subjects were included.

TMD diagnosis was based on the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD), following the 2014 Axis I protocol. Participants were classified into three groups:

None: No signs of TMD M: Muscular pain (myogenic) T: Joint-related pain (arthrogenic) The diagnostic process was based on clinical findings such as pain elicited by jaw movement, muscle palpation, or joint loading. Muscle-related pain was further subclassified according to whether the pain extended beyond anatomical boundaries (local muscle pain, myofascial pain, or referred pain). TMJ-originated pain was defined as pain induced by joint palpation or mandibular movements. TMJ-related headache diagnosis was based on pain elicited in the temporal area via palpation or functional movement.

Pain intensity and interference were assessed using the Graded Chronic Pain Scale Version 2.0 (GCPS v2.0). The Characteristic Pain Intensity (CPI) was calculated as the mean of items 2-4 multiplied by 10. The Interference Score was the mean of items 6-8, also multiplied by 10. Disability points were assigned based on the number of painful days in the past 30 days (item 5), resulting in a total pain grade from 0 (no pain) to 3 (severe pain).

Digital occlusal analysis was performed using the Medit i700 intraoral scanner (Medit Corp., Seoul, South Korea). All scans were taken once in the morning under maximum intercuspation. STL files were analyzed with the Medit Occlusal Analyzer plugin. Occlusal contact area percentages for premolars and molars were calculated, and non-contacting teeth were excluded. The average occlusal contact area per individual was used for statistical evaluation.

Tooth wear classification was performed using the Tooth Wear Evaluation System 2.0 (TWES 2.0) as proposed by Wetselaar et al. Occlusal/incisal and non-occlusal/non-incisal surfaces were graded on a 5-point ordinal scale.

For occlusal/incisal surfaces:

Grade 0: No visible wear Grade 1: Wear within enamel Grade 2: Dentin exposure with ≤1/3 crown height loss Grade 3: Crown height loss >1/3 but <2/3 Grade 4: Crown height loss ≥2/3

For non-occlusal surfaces (oral/vestibular):

Grade 0: No visible wear Grade 1: Wear within enamel Grade 2: Dentin exposure <50% of surface Grade 3: Dentin exposure ≥50% of surface Grade 4: Dentin exposure with total enamel/pulp loss Tooth wear grades were recorded separately for each tooth and surface. For statistical analysis, wear severity was simplified into three categories: no wear, enamel-level wear, and dentin-level wear.

Standardization and blinding were maintained by ensuring all scans and measurements were conducted by the same experienced prosthodontist using the same equipment in a controlled setting. TMD classification, wear evaluation, and pain assessment were carried out independently by different examiners.

Statistical analysis was performed using IBM SPSS Statistics 23. Shapiro-Wilk test assessed the normality of continuous variables. Non-parametric tests were used for non-normally distributed variables. Kruskal-Wallis test and Dwass-Steel-Critchlow-Fligner (DSCF) post hoc test with Bonferroni correction were used for group comparisons. Spearman's rho correlation was used to examine associations between variables. Multinomial logistic regression was applied to identify factors affecting TMD group classification. Ordinal logistic regression assessed the effects of pain level, wear severity, and occlusal contact. The interaction between pain and wear severity on TMD classification was analyzed using Generalized Linear Models (GLM). Statistical significance was set at p < 0.05.

Study limitations include its single-center design, limiting generalizability. Functional occlusal contacts during dynamic movements were not evaluated, and only static intercuspal position was analyzed. Additionally, due to insufficient data in pain Grade 4, this subgroup was excluded from analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above
* Voluntary participation with signed informed consent
* Presence of a sufficient number of posterior teeth (premolars and molars)
* Willingness to undergo intraoral digital scanning
* Willingness to participate in occlusal contact analysis procedures

Exclusion Criteria:

* Presence of systemic diseases affecting the temporomandibular joint (TMJ)
* Active dental pain at the time of evaluation
* Recent trauma to the facial or jaw region
* Current psychiatric or neurological disorders
* History of orthodontic treatment or extensive prosthetic rehabilitation
* Pathological jaw dysfunctions not related to parafunctional activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes individuals aged 18 years and older who have an adequate number of premolar and molar teeth in the posterior region, without systemic diseases, and without active dental pain or recent trauma to the face or neck. All participants were voluntarily selected from among patients who applied to the Department of Prosthodontics at the Faculty of Dentistry, Necmettin Erbakan University.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-12-26 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Occlusal contact area percentage in posterior teeth (%) | Baseline (Day 1 of clinical evaluation)
  Occlusal contact area will be calculated as a percentage of the total occlusal surface area in posterior teeth. Digital impressions will be acquired using the Medit i700 intraoral scanner. Contact points will be identified with the Medit Occlusal Analyzer plugin, and contact areas will be measured from STL files using ImageJ software (version 1.54). The percentage will be computed by dividing the total occlusal contact area by the total occlusal surface area.

SECONDARY OUTCOMES:
Tooth wear severity score assessed by TWES 2.0 (ordinal scale: 0-4) | Baseline (Day 1 of clinical evaluation)
  Tooth wear severity will be assessed visually according to the Tooth Wear Evaluation System 2.0 (TWES 2.0). Both occlusal/incisal and non-occlusal/non-incisal surfaces will be scored on a 0 to 4 ordinal scale. A composite severity score will be recorded for each participant.
Pain severity score using Graded Chronic Pain Scale v2.0 (unit: 0-4 categorical score) | Baseline (Day 1 of clinical evaluation)
  Pain severity will be assessed using the Graded Chronic Pain Scale version 2.0 (GCPS v2.0). The total score is derived by combining the Characteristic Pain Intensity (CPI), the disability score (based on the number of days with pain), and the functional interference score. The final score categorizes individuals into one of five levels (0 to 4), where higher scores indicate more severe and functionally limiting pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided